CLINICAL TRIAL: NCT01602120
Title: A Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of Lampalizumab (FCFD4514S) in Patients With Geographic Atrophy Who Have Completed Genentech-Sponsored Lampalizumab Studies
Brief Title: An Extension Study to Evaluate the Long-Term Safety of Lampalizumab in Participants With Geographic Atrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early by the Sponsor due to lack of efficacy.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX28198; 2012-000578-41 (EudraCT Number)
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — lampalizumab

ARMS (4):
- CFD4870g Sham (Experimental): Participants who were administered sham comparator in Study NCT01229215 (CFD4870g), will receive lampalizumab 10 milligrams (mg), intravitreally (ITV), either once in every 4 weeks (Q4W) or once in every 8 weeks (Q8W) in accordance with their previously assigned treatment frequency assignment in Study CFD4870g followed by Q4W administration for the remainder of the extension study up to approximately 96 months.
  Interventions: Drug: Lampalizumab
- CFD4870g Lampalizumab (Experimental): Participants will receive lampalizumab 10 mg, ITV, Q4W or Q8W in accordance with their previously assigned treatment frequency assignment in Study NCT01229215 (CFD4870g) followed by Q4W administration for the remainder of the extension study up to approximately 96 months.
  Interventions: Drug: Lampalizumab
- GX29455 Sham (Experimental): Participants who were administered sham comparator in Study NCT02288559 (GX29455), will receive lampalizumab 10 mg, ITV, Q4W throughout the extension study up to approximately 54 months.
  Interventions: Drug: Lampalizumab
- GX29455 Lampalizumab (Experimental): Participants who were administered lampalizumab in Study NCT02288559 (GX29455), will receive lampalizumab 10 mg, ITV, Q4W throughout the extension study up to approximately 54 months.
  Interventions: Drug: Lampalizumab

INTERVENTIONS:
Drug: Lampalizumab — Lampalizumab 10 mg ITV injections as per the schedule specified in respective arms.
  Other Names: FCFD4514S

SUMMARY:
This is a multicenter, open-label extension study of safety and tolerability of lampalizumab administered by intravitreal (ITV) injection to participants with geographic atrophy (GA) who have completed the 18-month treatment in Study CFD4870g (GX01456) (NCT01229215) or 24-week treatment in Study GX29455 (NCT02288559).

ELIGIBILITY:
Inclusion Criteria:

* For CFD4870g participants: Previous enrollment and completion (Month 18 visit) of Study CFD4870g without early treatment discontinuation (lampalizumab or sham)
* For GX29455 participants: Previous enrollment and completion (Week 24 visit) of Study GX29455 without early treatment discontinuation (lampalizumab or sham)
* Sufficiently clear ocular media, adequate pupillary dilation, and fixation to permit quality fundus imaging

Exclusion Criteria:

* Early treatment and/or study discontinuation prior to completion of study CFD4870g (GX01456) and GX29455
* Vitrectomy surgery, submacular surgery, or other surgical intervention for age-related macular degeneration (AMD) in the study eye
* Subfoveal focal laser photocoagulation in the study eye
* Treatment with Visodyne, external-beam radiation therapy, or transpupillary thermotherapy in the study eye
* Intravitreally (ITV) drug delivery (e.g., ITV corticosteroid injection, anti-angiogenic drugs, anticomplement drugs, or device implantation) in the study eye. Lampalizumab in study eye and ranibizumab in either eye are permitted
* Any concurrent ocular or intraocular condition in the study eye that contraindicates the use of an investigational drug or may affect interpretation of the study results or may render the participant at high risk for treatment complications

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (46):
- United States (41):
  - Retina Centers P.C., Tucson, Arizona
  - Retina-Vitreous Assoc Med Grp, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - Loma Linda University, Loma Linda, California
  - San Diego Retina Associates, Oceanside, California
  - W Coast Retina Med Group Inc, San Francisco, California
  - West Coast Retina, San Francisco, California
  - California Retina Consultants, Santa Barbara, California
  - Retina Macula Institute, Torrance, California
  - Colorado Retina Associates, PC, Golden, Colorado
  - Retina Group of Florida, Boca Raton, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Ctr for Retina & Macular Dis, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Elman Retina Group, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreoretinal Surgery, Edina, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Opthalmic Consultants of LI, Lynbrook, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Retina Assoc of Cleveland Inc, Beachwood, Ohio
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Northwest, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - W Texas Retina Consultants PA, Abilene, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Wagner Macula & Retina Center, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (5):
  - Universitatsklinikum Bonn; Medizinische Klinik und Poliklinik III, Bonn
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Leipzig, Leipzig
  - St. Franziskus Hospital, Münster
  - Universitätsklinikum Tübingen, Tübingen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled eligible patients who had completed the 18-month treatment period of Study NCT01229215 (CFD4870g) or the 24-week treatment period of Study NCT02288559 (GX29455). The study was terminated early by the Sponsor due to lack of efficacy.
Groups:
- CFD4870g Sham: Participants who were administered sham comparator in Study NCT01229215 (CFD4870g), received lampalizumab 10 milligrams (mg), intravitreally (ITV), either once in every 4 weeks (Q4W) or once in every 8 weeks (Q8W) in accordance with their previously assigned treatment frequency assignment in Study CFD4870g followed by Q4W administration for the remainder of the extension study.
- CFD4870g Lampalizumab: Participants received lampalizumab 10 mg, ITV, Q4W or Q8W in accordance with their previously assigned treatment frequency assignment in Study NCT01229215 (CFD4870g) followed by Q4W administration for the remainder of the extension study.
- GX29455 Sham: Participants who were administered sham comparator in Study NCT02288559 (GX29455), received lampalizumab 10 mg, ITV, Q4W throughout the extension study.
- GX29455 Lampalizumab: Participants who were administered lampalizumab in Study NCT02288559 (GX29455), received lampalizumab 10 mg, ITV, Q4W throughout the extension study.
Period: Overall Study
Arm/Group | CFD4870g Sham | CFD4870g Lampalizumab | GX29455 Sham | GX29455 Lampalizumab
Started | 29 | 60 | 17 | 53
Completed | 0 | 0 | 0 | 0
Not Completed | 29 | 60 | 17 | 53
Not completed — Adverse Event | 3 | 6 | 0 | 2
Not completed — Death | 0 | 4 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 17 | 0 | 3
Not completed — Study Terminated by Sponsor | 12 | 24 | 17 | 44
Not completed — Physician Decision | 2 | 3 | 0 | 0
Not completed — Unspecified Reason | 3 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled and received at least one lampalizumab injection in the extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | CFD4870g Sham | CFD4870g Lampalizumab | GX29455 Sham | GX29455 Lampalizumab | Total
Number analyzed (Participants) | 29 | 60 | 17 | 53 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.4 (6.6) | 79.4 (6.8) | 76.7 (6.6) | 79.5 (7.6) | 79.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 33 | 12 | 27 | 89
  Male | 12 | 27 | 5 | 26 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 29 | 59 | 17 | 52 | 157
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 29 | 59 | 15 | 53 | 156

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ocular and Non-ocular Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, or any deterioration in a laboratory value or other clinical test. Ocular AEs are events localized to the eye. Non-ocular events include all other events.
Time Frame: From Day 1 up to the last study visit (up to approximately 62 months)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- All Participants: All participants in the study received lampalizumab 10 mg, ITV, Q4W.
Arm/Group | CFD4870g Sham | CFD4870g Lampalizumab | GX29455 Sham | GX29455 Lampalizumab | All Participants
Number analyzed (Participants) | 29 | 60 | 17 | 53 | 159
percentage of participants
  Ocular AEs in Study Eye | 62.1 | 78.3 | 52.9 | 50.9 | 63.5
  Ocular AEs in Fellow Eye | 62.1 | 68.3 | 29.4 | 60.4 | 60.4
  Non-Ocular AEs | 79.3 | 90.0 | 82.4 | 67.9 | 79.9

ADVERSE EVENTS:
Time Frame: From Day 1 up to the last study visit (up to approximately 62 months)
Description: At the time of study enrollment, if the participant had any ongoing adverse events from Study NCT01229215 (CFD4870g) or NCT02288559 (GX29455) these events were counted in this study. Safety population included all participants who were enrolled and received at least one lampalizumab injection in the extension study. The arm All Participants reports all adverse events that occurred in the four arms in the study.
Arm/Group | CFD4870g Sham | CFD4870g Lampalizumab | GX29455 Sham | GX29455 Lampalizumab | All Participants
All-Cause Mortality (participants affected / at risk) | 1/29 | 6/60 | 0/17 | 1/53 | 8/159
Serious Adverse Events (participants affected / at risk) | 16/29 | 40/60 | 5/17 | 9/53 | 70/159
Other Adverse Events (participants affected / at risk) | 24/29 | 56/60 | 16/17 | 41/53 | 137/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFD4870g Sham (N=29) | CFD4870g Lampalizumab (N=60) | GX29455 Sham (N=17) | GX29455 Lampalizumab (N=53) | All Participants (N=159)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 1 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 5 | 0 | 0 | 5
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 4 | 0 | 0 | 4
Cardiac perforation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2 | 0 | 0 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 2 | 0 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Ventricle rupture (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Blindness transient (Eye disorders) | 0 | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 2 | 2 | 1 | 0 | 5
Visual impairment (Eye disorders) | 0 | 2 | 0 | 0 | 2
Vitritis (Eye disorders) | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2 | 0 | 0 | 4
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Infected lymphocele (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 4 | 0 | 1 | 6
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Genital injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 2
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CFD4870g Sham (N=29) | CFD4870g Lampalizumab (N=60) | GX29455 Sham (N=17) | GX29455 Lampalizumab (N=53) | All Participants (N=159)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 10 | 1 | 2 | 15
Coronary artery disease (Cardiac disorders) | 1 | 4 | 0 | 0 | 5
Cardiac failure congestive (Cardiac disorders) | 0 | 3 | 0 | 1 | 4
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 4 | 18 | 3 | 3 | 28
Retinal haemorrhage (Eye disorders) | 4 | 13 | 2 | 3 | 22
Eye pain (Eye disorders) | 3 | 14 | 0 | 4 | 21
Cataract (Eye disorders) | 1 | 9 | 0 | 5 | 15
Posterior capsule opacification (Eye disorders) | 3 | 3 | 2 | 5 | 13
Vitreous detachment (Eye disorders) | 4 | 2 | 0 | 6 | 12
Vitreous floaters (Eye disorders) | 2 | 6 | 1 | 3 | 12
Dry eye (Eye disorders) | 1 | 6 | 0 | 4 | 11
Punctate keratitis (Eye disorders) | 1 | 7 | 2 | 1 | 11
Visual impairment (Eye disorders) | 0 | 5 | 1 | 3 | 9
Cataract nuclear (Eye disorders) | 1 | 3 | 0 | 4 | 8
Blepharitis (Eye disorders) | 1 | 4 | 0 | 2 | 7
Neovascular age-related macular degeneration (Eye disorders) | 2 | 3 | 1 | 1 | 7
Vision blurred (Eye disorders) | 3 | 4 | 0 | 0 | 7
Iritis (Eye disorders) | 1 | 4 | 1 | 0 | 6
Blindness transient (Eye disorders) | 1 | 4 | 0 | 0 | 5
Cataract subcapsular (Eye disorders) | 0 | 4 | 1 | 0 | 5
Dry age-related macular degeneration (Eye disorders) | 2 | 2 | 0 | 1 | 5
Eye pruritus (Eye disorders) | 1 | 3 | 1 | 0 | 5
Lacrimation increased (Eye disorders) | 2 | 1 | 0 | 2 | 5
Ocular hyperaemia (Eye disorders) | 1 | 3 | 0 | 1 | 5
Foreign body sensation in eyes (Eye disorders) | 1 | 3 | 0 | 0 | 4
Visual acuity reduced (Eye disorders) | 2 | 1 | 0 | 1 | 4
Blepharochalasis (Eye disorders) | 0 | 0 | 0 | 3 | 3
Conjunctival hyperaemia (Eye disorders) | 2 | 1 | 0 | 0 | 3
Ocular hypertension (Eye disorders) | 0 | 0 | 0 | 3 | 3
Open angle glaucoma (Eye disorders) | 1 | 0 | 1 | 1 | 3
Trichiasis (Eye disorders) | 2 | 1 | 0 | 0 | 3
Corneal erosion (Eye disorders) | 2 | 0 | 0 | 0 | 2
Corneal opacity (Eye disorders) | 0 | 1 | 1 | 0 | 2
Vitreous haemorrhage (Eye disorders) | 2 | 0 | 0 | 0 | 2
Corneal oedema (Eye disorders) | 0 | 0 | 1 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 1 | 0 | 1
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 9 | 1 | 1 | 13
Diarrhoea (Gastrointestinal disorders) | 1 | 7 | 0 | 2 | 10
Nausea (Gastrointestinal disorders) | 1 | 5 | 0 | 2 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 5 | 0 | 0 | 7
Gastritis (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 5
Oedema peripheral (General disorders) | 2 | 3 | 1 | 2 | 8
Pain (General disorders) | 1 | 3 | 0 | 0 | 4
Asthenia (General disorders) | 0 | 3 | 0 | 0 | 3
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 3 | 0 | 0 | 4
Drug hypersensitivity (Immune system disorders) | 0 | 3 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 8 | 11 | 1 | 4 | 24
Urinary tract infection (Infections and infestations) | 3 | 13 | 1 | 4 | 21
Upper respiratory tract infection (Infections and infestations) | 4 | 9 | 3 | 4 | 20
Bronchitis (Infections and infestations) | 5 | 7 | 0 | 2 | 14
Sinusitis (Infections and infestations) | 4 | 5 | 1 | 1 | 11
Pneumonia (Infections and infestations) | 0 | 6 | 1 | 2 | 9
Herpes zoster (Infections and infestations) | 1 | 4 | 0 | 2 | 7
Influenza (Infections and infestations) | 0 | 6 | 1 | 0 | 7
Cystitis (Infections and infestations) | 1 | 3 | 0 | 1 | 5
Ear infection (Infections and infestations) | 0 | 4 | 1 | 0 | 5
Conjunctivitis (Infections and infestations) | 1 | 3 | 0 | 0 | 4
Tooth infection (Infections and infestations) | 1 | 3 | 0 | 0 | 4
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0 | 3
Diverticulitis (Infections and infestations) | 0 | 3 | 0 | 0 | 3
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 7 | 13 | 3 | 2 | 25
Contusion (Injury, poisoning and procedural complications) | 0 | 5 | 0 | 1 | 6
Procedural pain (Injury, poisoning and procedural complications) | 1 | 5 | 0 | 0 | 6
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 0 | 5
Laceration (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 4
Rib fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0 | 4
Muscle strain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Intraocular pressure increased (Investigations) | 3 | 6 | 0 | 3 | 12
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 1 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 2 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 2 | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 0 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1 | 6
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 5
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 3
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 0 | 6
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 3
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 3
Headache (Nervous system disorders) | 1 | 8 | 0 | 0 | 9
Dementia (Nervous system disorders) | 1 | 3 | 0 | 1 | 5
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 1 | 4
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 1 | 0 | 4
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 4 | 0 | 1 | 6
Anxiety (Psychiatric disorders) | 0 | 3 | 0 | 2 | 5
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 1 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 4 | 0 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 1 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 3
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2
Cataract operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 7 | 1 | 1 | 11
Hypotension (Vascular disorders) | 0 | 4 | 1 | 0 | 5
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor, because the compound had demonstrated lack of efficacy. Thus, no participant in this study completed the full duration of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT01602120/Prot_SAP_000.pdf